CLINICAL TRIAL: NCT01652885
Title: An Open-Label Study to Determine the Safety, Tolerability, and Pharmacokinetic Profile of AN2728 Ointment in Adolescents With Atopic Dermatitis
Brief Title: Safety, Tolerability, and PK of AN2728 in Adolescents With Atopic Dermatitis
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AN2728-AD-203; A3191007 (Other: Pfizer)
Record Dates: First submitted 2012-07-20; First posted 2012-07-30 (Estimated); Results first posted 2017-04-24 (Actual); Last update posted 2017-04-24 (Actual); Status verified 2017-03

CONDITIONS: Dermatitis, Atopic
Keywords: atopic dermatitis
MeSH Terms: conditions — Dermatitis, Atopic

ARMS (1):
- AN2728 Topical Ointment, 2% (Experimental): AN2728 Topical Ointment, 2%, applied twice daily for up to 28 days
  Interventions: Drug: AN2728 Topical Ointment, 2%

INTERVENTIONS:
Drug: AN2728 Topical Ointment, 2% — AN2728 Topical Ointment, 2%

SUMMARY:
The purpose of this study is to investigate the safety, tolerability, and systemic exposure of AN2728 Topical Ointment, 2%, in subjects with atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female 12 to 17 years of age, inclusive
* Clinical diagnosis of atopic dermatitis (according to the criteria of Hanifin and Rajka)
* AD in treatable areas (excludes the scalp and venous access areas) involving

  ≥10% and ≤35% of the total body surface area(BSA)
* Investigator's Static Global Assessment (ISGA) score of 2 or 3
* Normal or not clinically significant screening laboratory results
* Have adequate venous access to permit repeated PK sampling on Days 1 - 9 through uninfected skin that has not been treated with study drug; each untreated venous access area should provide a margin of at least 5 cm radius around the venipuncture site
* Willing and able to comply with study instructions and commit to attending all visits
* Females must use a highly effective method of birth control.
* Parent/guardian has the ability to understand, agree to and sign the study Informed Consent Form (ICF) prior to initiation of any protocol-related procedures; subject has the ability to give assent

Exclusion Criteria:

* Significant confounding conditions as assessed by study doctor
* Unstable or actively infected AD
* Active or potentially recurrent dermatologic condition other than atopic dermatitis that may confound evaluation
* History or evidence of allergies requiring acute or chronic treatment (except seasonal allergic rhinitis)
* Concurrent or recent use of certain topical or systemic medications or phototherapy without a sufficient washout period
* Treatment for any type of cancer (except squamous cell carcinoma, basal cell carcinoma, or carcinoma in situ of the skin, curatively treated with cryosurgery or surgical excision only) within the last 5 years
* Current pregnancy or lactation, or intent to become pregnant during the study
* Known sensitivity to any of the components of the study drug
* Participated in any other trial of an investigational drug or device within 30 days or participation in a research study concurrent with this study
* Participated in a previous AN2728 clinical study

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 23 (Actual)
Dates: Start 2012-07; Primary Completion 2012-10 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (6):
- United States (6):
  - Anacor Investigational Site, Fremont, California
  - Anacor Investigational Site, San Diego, California
  - Anacor Investigational Site, Indianapolis, Indiana
  - Anacor Investigational Site, High Point, North Carolina
  - Anacor Investigational Site, Winston-Salem, North Carolina
  - Anacor Investigational Site, Houston, Texas

RESULTS

PARTICIPANT FLOW:
Groups:
- AN2728 Topical Ointment 2 Percent: AN2728 ointment 2 percent was applied topically to treatment-targeted lesions in participant with mild to moderate atopic dermatitis (AD), twice daily for up to 28 days, except on Day 1 and 8 applied once daily. Lesions were identified at Baseline (Day 1) by investigator.
Period: Overall Study
Arm/Group | AN2728 Topical Ointment 2 Percent
Started | 23
Completed | 22
Not Completed | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Population: Safety population included all participants who were enrolled and had received any amount of study drug.
Groups:
- AN2728 Topical Ointment 2 Percent: AN2728 ointment 2 percent was applied topically to treatment-targeted lesions in participant with mild to moderate AD, twice daily for up to 28 days, except on Day 1 and 8 applied once daily. Lesions were identified at Baseline (Day 1) by investigator.
Arm/Group | AN2728 Topical Ointment 2 Percent
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 15.0 (1.55)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 4

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Local Tolerability Symptoms According to Severity on Baseline
Description: Local tolerability symptoms, burning or stinging, were classified according to severity as: 1) none = no stinging or burning, 2) mild = slight warm, tingling sensation; not really troublesome, 3) moderate = definite warm; tingling or stinging sensation; troublesome and 4) severe = hot, tingling or stinging sensation that caused definite discomfort. Number of participants with local tolerability symptoms according to severity on Baseline were reported in this outcome measure.
Time Frame: Baseline
Population: Safety population included all participants who were enrolled and had received any amount of the study drug.
Measure: Number; unit: participants
Arm/Group | AN2728 Topical Ointment 2 Percent
Number analyzed (Participants) | 23
participants
  None | 10
  Mild | 7
  Moderate | 6
  Severe | 0

2. Primary Outcome: Number of Participants With Local Tolerability Symptoms According to Severity on Day 2
Description: Local tolerability symptoms, burning or stinging, were classified according to severity as: 1) none = no stinging or burning, 2) mild = slight warm, tingling sensation; not really troublesome, 3) moderate = definite warm; tingling or stinging sensation; troublesome and 4) severe = hot, tingling or stinging sensation that caused definite discomfort. Number of participants with local tolerability symptoms according to severity on Day 2 were reported in this outcome measure.
Time Frame: Day 2
Population: Safety population included all participants who were enrolled and had received any amount of the study drug.
Measure: Number; unit: participants
Arm/Group | AN2728 Topical Ointment 2 Percent
Number analyzed (Participants) | 23
participants
  None | 17
  Mild | 5
  Moderate | 1
  Severe | 0

3. Primary Outcome: Number of Participants With Local Tolerability Symptoms According to Severity on Day 4
Description: Local tolerability symptoms, burning or stinging, were classified according to severity as: 1) none = no stinging or burning, 2) mild = slight warm, tingling sensation; not really troublesome, 3) moderate = definite warm; tingling or stinging sensation; troublesome and 4) severe = hot, tingling or stinging sensation that caused definite discomfort. Number of participants with local tolerability symptoms according to severity on Day 4 were reported in this outcome measure.
Time Frame: Day 4
Population: Safety population included all participants who were enrolled and had received any amount of the study drug.
Measure: Number; unit: participants
Arm/Group | AN2728 Topical Ointment 2 Percent
Number analyzed (Participants) | 23
participants
  None | 18
  Mild | 3
  Moderate | 2
  Severe | 0

4. Primary Outcome: Number of Participants With Local Tolerability Symptoms According to Severity on Day 6
Description: Local tolerability symptoms, burning or stinging, were classified according to severity as: 1) none = no stinging or burning, 2) mild = slight warm, tingling sensation; not really troublesome, 3) moderate = definite warm; tingling or stinging sensation; troublesome and 4) severe = hot, tingling or stinging sensation that caused definite discomfort. Number of participants with local tolerability symptoms according to severity on Day 6 were reported in this outcome measure.
Time Frame: Day 6
Population: Safety population included all participants who were enrolled and had received any amount of the study drug.
Measure: Number; unit: participants
Arm/Group | AN2728 Topical Ointment 2 Percent
Number analyzed (Participants) | 23
participants
  None | 18
  Mild | 4
  Moderate | 1
  Severe | 0

5. Primary Outcome: Number of Participants With Local Tolerability Symptoms According to Severity on Day 8
Description: Local tolerability symptoms, burning or stinging, were classified according to severity as: 1) none = no stinging or burning, 2) mild = slight warm, tingling sensation; not really troublesome, 3) moderate = definite warm; tingling or stinging sensation; troublesome and 4) severe = hot, tingling or stinging sensation that caused definite discomfort. Number of participants with local tolerability symptoms according to severity on Day 8 were reported in this outcome measure.
Time Frame: Day 8
Population: Safety population included all participants who were enrolled and had received any amount of the study drug.
Measure: Number; unit: participants
Arm/Group | AN2728 Topical Ointment 2 Percent
Number analyzed (Participants) | 23
participants
  None | 20
  Mild | 3
  Moderate | 0
  Severe | 0

6. Primary Outcome: Number of Participants With Local Tolerability Symptoms According to Severity on Day 9
Description: Local tolerability symptoms, burning or stinging, were classified according to severity as: 1) none = no stinging or burning, 2) mild = slight warm, tingling sensation; not really troublesome, 3) moderate = definite warm; tingling or stinging sensation; troublesome and 4) severe = hot, tingling or stinging sensation that caused definite discomfort. Number of participants with local tolerability symptoms according to severity on Day 9 were reported in this outcome measure.
Time Frame: Day 9
Population: Safety population included all participants who were enrolled and had received any amount of the study drug.
Measure: Number; unit: participants
Arm/Group | AN2728 Topical Ointment 2 Percent
Number analyzed (Participants) | 23
participants
  None | 18
  Mild | 4
  Moderate | 1
  Severe | 0

7. Primary Outcome: Number of Participants With Local Tolerability Symptoms According to Severity on Day 15
Description: Local tolerability symptoms, burning or stinging, were classified according to severity as: 1) none = no stinging or burning, 2) mild = slight warm, tingling sensation; not really troublesome, 3) moderate = definite warm; tingling or stinging sensation; troublesome and 4) severe = hot, tingling or stinging sensation that caused definite discomfort. Number of participants with local tolerability symptoms according to severity on Day 15 were reported in this outcome measure.
Time Frame: Day 15
Population: Safety population included all participants who were enrolled and had received any amount of the study drug.
Measure: Number; unit: participants
Arm/Group | AN2728 Topical Ointment 2 Percent
Number analyzed (Participants) | 23
participants
  None | 19
  Mild | 4
  Moderate | 0
  Severe | 0

8. Primary Outcome: Number of Participants With Local Tolerability Symptoms According to Severity on Day 22
Description: Local tolerability symptoms, burning or stinging, were classified according to severity as: 1) none = no stinging or burning, 2) mild = slight warm, tingling sensation; not really troublesome, 3) moderate = definite warm; tingling or stinging sensation; troublesome and 4) severe = hot, tingling or stinging sensation that caused definite discomfort. Number of participants with local tolerability symptoms according to severity on Day 22 were reported in this outcome measure.
Time Frame: Day 22
Population: Safety population included all participants who were enrolled and had received any amount of the study drug.
Measure: Number; unit: participants
Arm/Group | AN2728 Topical Ointment 2 Percent
Number analyzed (Participants) | 23
participants
  None | 21
  Mild | 2
  Moderate | 0
  Severe | 0

9. Primary Outcome: Number of Participants With Local Tolerability Symptoms According to Severity on Day 29
Description: Local tolerability symptoms, burning or stinging, were classified according to severity as: 1) none = no stinging or burning, 2) mild = slight warm, tingling sensation; not really troublesome, 3) moderate = definite warm; tingling or stinging sensation; troublesome and 4) severe = hot, tingling or stinging sensation that caused definite discomfort. Number of participants with local tolerability symptoms according to severity on Day 29 were reported in this outcome measure.
Time Frame: Day 29
Population: Safety population included all participants who were enrolled and had received any amount of the study drug.
Measure: Number; unit: participants
Arm/Group | AN2728 Topical Ointment 2 Percent
Number analyzed (Participants) | 23
participants
  None | 20
  Mild | 2
  Moderate | 0
  Severe | 1

10. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. An SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death;initial or prolonged inpatient hospitalization; life- threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. Treatment-emergent were events between first dose of study drug and up to Day 29 that were absent before treatment or that worsened relative to pretreatment state.
Time Frame: Baseline (Day 1) up to Day 29
Population: Safety population included all participants who were enrolled and had received any amount of the study drug.
Measure: Number; unit: participants
Arm/Group | AN2728 Topical Ointment 2 Percent
Number analyzed (Participants) | 23
participants
  AEs | 10
  SAEs | 0

11. Primary Outcome: Number of Participants With Clinically Significant Vital Signs Abnormalities
Description: Vital signs (temperature, respiratory rate, pulse, systolic and diastolic blood pressure) were obtained with participant in the seated position, after having sat calmly for at least 5 minutes. Clinical significance of vital signs was determined at the investigator's discretion.
Time Frame: Baseline (Day 1) up to Day 29
Population: Safety population included all participants who were enrolled and had received any amount of the study drug.
Measure: Number; unit: participants
Arm/Group | AN2728 Topical Ointment 2 Percent
Number analyzed (Participants) | 23
participants | 0

12. Primary Outcome: Number of Participants With Clinically Significant Laboratory Test Abnormalities
Description: Laboratory parameters included: hematology (hemoglobin, hematocrit, red blood cell, platelet and white blood cell count, neutrophils, eosinophils, monocytes, basophils and lymphocytes), chemistry (blood urea nitrogen, creatinine, sodium, potassium, aspartate aminotransferase, alanine aminotransferase, total bilirubin, alkaline phosphatase, albumin, total protein and serum pregnancy test [for all female participants]) and urine (urine pregnancy test [for all female participants]). Clinical significance of laboratory parameters was determined at the investigator's discretion.
Time Frame: Baseline (Day 1) up to Day 29
Population: Safety population included all participants who were enrolled and had received any amount of the study drug.
Measure: Number; unit: participants
Arm/Group | AN2728 Topical Ointment 2 Percent
Number analyzed (Participants) | 23
participants | 0

13. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of AN2728 and Major Oxidative Metabolites of AN2728: Day 1
Description: Maximum observed plasma concentration of AN2728 and its two identified oxidative metabolites, AN7602 and AN8323 on Day 1 was reported in the outcome measure.
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 8, 12 and 24 hours post-dose on Day 1
Population: Pharmacokinetic (PK) population included participants from the safety population who had completed any portion of the PK day procedures and evaluations.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | AN2728 Topical Ointment 2 Percent
Number analyzed (Participants) | 23
nanogram per milliliter
  AN2728 | 105 (160)
  AN7602 | 28.2 (37.0)
  AN8323 | 998 (1220)

14. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of AN2728 and Major Oxidative Metabolites of AN2728: Day 1
Description: Time to reach maximum plasma concentration of AN2728 and its two identified oxidative metabolites, AN7602 and AN8323 on Day 1 was reported in the outcome measure.
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 8, 12 and 24 hours post-dose on Day 1
Population: PK population included participants from the safety population who had completed any portion of the PK day procedures and evaluations.
Measure: Median (Full Range); unit: hour
Arm/Group | AN2728 Topical Ointment 2 Percent
Number analyzed (Participants) | 23
hour
  AN2728 | 2.37 [1.00 to 24.0]
  AN7602 | 2.08 [1.00 to 24.0]
  AN8323 | 6.25 [3.95 to 25.0]

15. Primary Outcome: Area Under the Concentration-Time Curve From Hour Zero To the 12 Hour Post-Dose Measurable Concentration of AN2728 and Major Oxidative Metabolites of AN2728: Day 1
Description: Area under the concentration-time curve from hour zero to the 12 hour post-dose measurable concentration, of AN2728 and its two identified oxidative metabolites, AN7602 and AN8323 on Day 1 was reported in the outcome measure.
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 8 and 12 hours post-dose on Day 1
Population: as for outcome 14
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter
Arm/Group | AN2728 Topical Ointment 2 Percent
Number analyzed (Participants) | 23
nanogram*hour per milliliter
  AN2728 | 448 (527)
  AN7602 | 142 (172)
  AN8323 | 8900 (11600)

16. Primary Outcome: Apparent Terminal Half-Life of AN2728 and Major Oxidative Metabolites of AN2728: Day 1
Description: Apparent terminal half-life, of AN2728 and its two identified oxidative metabolites, AN7602 and AN8323 on Day 1 was reported in the outcome measure. Apparent terminal half-life is the time measured for the drug concentration to decrease by one-half in plasma.
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 8, 12 and 24 hours post-dose on Day 1
Population: PK population included participants from the safety population who had completed any portion of the PK day procedures and evaluations. Here, "n" signifies number of participants who were evaluable for specific categories.
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | AN2728 Topical Ointment 2 Percent
Number analyzed (Participants) | 23
hour
  AN2728 (n =16) | 7.17 (2.30)
  AN7602 (n =18) | 8.19 (5.13)
  AN8323 (n =6) | 17.7 (1.63)

17. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of AN2728 and Major Oxidative Metabolites of AN2728: Day 8
Description: Maximum observed plasma concentration of AN2728 and its two identified oxidative metabolites, AN7602 and AN8323 on Day 8 was reported in the outcome measure.
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 8, 12 and 24 hours post-dose on Day 8
Population: PK population included participants from the safety population who had completed any portion of the PK day procedures and evaluations. Here, "Number of Participants Analyzed" (N) signifies evaluable participants for this outcome measure.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter
Arm/Group | AN2728 Topical Ointment 2 Percent
Number analyzed (Participants) | 22
nanogram per milliliter
  AN2728 | 94.6 (189)
  AN7602 | 26.3 (43.9)
  AN8323 | 1850 (1830)

18. Primary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax) of AN2728 and Major Oxidative Metabolites of AN2728: Day 8
Description: Time to reach maximum plasma concentration of AN2728 and its two identified oxidative metabolites, AN7602 and AN8323 on Day 8 was reported in the outcome measure.
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 8, 12 and 24 hours post-dose on Day 8
Population: PK population included participants from the safety population who had completed any portion of the PK day procedures and evaluations. Here, 'N' signifies evaluable participants for this outcome measure.
Measure: Median (Full Range); unit: hour
Arm/Group | AN2728 Topical Ointment 2 Percent
Number analyzed (Participants) | 22
hour
  AN2728 | 2.17 [1.00 to 7.93]
  AN7602 | 3.94 [1.00 to 6.15]
  AN8323 | 6.00 [0.00 to 25.1]

19. Primary Outcome: Area Under the Concentration-Time Curve From Hour Zero To the 12 Hour Post-Dose Measurable Concentration of AN2728 and Major Oxidative Metabolites of AN2728: Day 8
Description: Area under the concentration-time curve from hour zero to the 12 hour post-dose measurable concentration, of AN2728 and its two identified oxidative metabolites, AN7602 and AN8323 on Day 8 was reported in the outcome measure.
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 8 and 12 hours post-dose on Day 8
Population: as for outcome 18
Measure: Mean (Standard Deviation); unit: nanogram*hour per milliliter
Arm/Group | AN2728 Topical Ointment 2 Percent
Number analyzed (Participants) | 22
nanogram*hour per milliliter
  AN2728 | 462 (506)
  AN7602 | 142 (154)
  AN8323 | 18200 (18100)

20. Primary Outcome: Apparent Terminal Half-Life of AN2728 and Major Oxidative Metabolites of AN2728: Day 8
Description: Apparent terminal half-life, of AN2728 and its two identified oxidative metabolites, AN7602 and AN8323 on Day 8 was reported in the outcome measure. Apparent terminal half-life is the time measured for the drug concentration to decrease by one-half in plasma.
Time Frame: Pre-dose (0 hour), 1, 2, 4, 6, 8, 12 and 24 hours post-dose on Day 8
Population: as for outcome 16
Measure: Mean (Standard Deviation); unit: hour
Arm/Group | AN2728 Topical Ointment 2 Percent
Number analyzed (Participants) | 23
hour
  AN2728 (n =17) | 11.9 (8.28)
  AN7602 (n =16) | 10.5 (6.38)
  AN8323 (n =6) | 33.5 (10.1)

21. Secondary Outcome: Number of Participants Who Achieved Treatment Success Based on Investigator's Static Global Assessment (ISGA)
Description: ISGA assess severity of atopic dermatitis on a 5 point scale ranged from 0 (clear) to 4 (maximum severe), where higher scores indicate higher degree of atopic dermatitis. Grades for classification of severity: 0= clear (minor residual discoloration, no erythema or induration or papulation, no oozing or crusting), 1= almost clear (trace faint pink erythema, with barely perceptible induration or papulation and no oozing or crusting), 2= mild (faint pink erythema with mild induration or papulation and no oozing or crusting), 3= moderate (pink-red erythema with moderate induration or papulation with or without oozing or crusting) and 4= severe (deep or bright red erythema with severe induration or papulation and with oozing or crusting). Treatment success was defined as ISGA score of 0 or 1, and a minimum improvement of 2 grades in ISGA from Baseline to Day 29.
Time Frame: Baseline up to Day 29
Population: Safety population included all participants who were enrolled and had received any amount of the study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | AN2728 Topical Ointment 2 Percent
Number analyzed (Participants) | 23
Participants | 9

22. Secondary Outcome: Change From Baseline in Signs and Symptoms of Atopic Dermatitis at Day 8, 15, 22 and 29
Description: 5 signs and symptoms of atopic dermatitis were: 1) erythema, 2) pruritus, 3) exudation, 4) excoriation and 5) lichenification. The severity of each of these 5 signs and symptoms were assessed on a 4 point scale, ranging from 0 (none) to 3 (severe). Higher scores (for each of the 5 signs and symptoms) indicate higher degree of severity of atopic dermatitis.
Time Frame: Baseline, Day 8, 15, 22, 29
Population: Safety population included all participants who were enrolled and had received any amount of the study drug.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | AN2728 Topical Ointment 2 Percent
Number analyzed (Participants) | 23
units on a scale
  Baseline: Erythema | 1.63 (0.607)
  Change at Day 8: Erythema | -0.63 (0.588)
  Change at Day 15: Erythema | -0.70 (0.617)
  Change at Day 22: Erythema | -0.87 (0.626)
  Change at Day 29: Erythema | -0.89 (0.673)
  Baseline: Pruritus | 1.87 (0.815)
  Change at Day 8: Pruritus | -1.11 (0.916)
  Change at Day 15: Pruritus | -1.11 (0.825)
  Change at Day 22: Pruritus | -1.15 (0.804)
  Change at Day 29: Pruritus | -1.30 (0.735)
  Baseline: Exudation | 0.33 (0.467)
  Change at Day 8: Exudation | -0.20 (0.328)
  Change at Day 15: Exudation | -0.20 (0.328)
  Change at Day 22: Exudation | -0.09 (0.492)
  Change at Day 29: Exudation | -0.07 (0.645)
  Baseline: Excoriation | 1.04 (0.689)
  Change at Day 8: Excoriation | -0.50 (0.603)
  Change at Day 15: Excoriation | -0.57 (0.728)
  Change at Day 22: Excoriation | -0.52 (0.805)
  Change at Day 29: Excoriation | -0.61 (0.852)
  Baseline: Lichenification | 1.67 (0.614)
  Change at Day 8: Lichenification | -0.54 (0.520)
  Change at Day 15: Lichenification | -0.59 (0.596)
  Change at Day 22: Lichenification | -0.85 (0.573)
  Change at Day 29: Lichenification | -0.78 (0.671)

ADVERSE EVENTS:
Arm/Group | AN2728 Topical Ointment 2 Percent
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 10/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | AN2728 Topical Ointment 2 Percent (N=23)
Application site dermatitis (General disorders) | 1
Application site discomfort (General disorders) | 1
Application site pain (General disorders) | 3
Upper respiratory tract infection (Infections and infestations) | 1
Arthropod bite (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Headache (Nervous system disorders) | 1
Migraine (Nervous system disorders) | 1
Dysmenorrhoea (Reproductive system and breast disorders) | 1/19 — This event was gender specific.
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 3
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 1
Milia (Skin and subcutaneous tissue disorders) | 1
Solar dermatitis (Skin and subcutaneous tissue disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.